CLINICAL TRIAL: NCT06617611
Title: What Matters to You on the Day of Surgery 2024?
Acronym: WMTY2024
Status: Completed | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Brigitta Rasmussen Villumsen, Postdoc, Gødstrup Hospital
Other Study IDs: 1-16-02-118-24
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Surgical Fear and Worrying; Person-centered Care
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgical intervention and anesthesia — Any surgical procedure

SUMMARY:
Research show that between 48-97% of patients referred to surgery experience anxiety and fear related to the procedure. High levels of anxiety and fear lead to increased use of anesthetics and pain as well as increased morbidity after the surgical procedure.

June 6 2024 is the international "What matters to you-day" and thus we mark this day in several Danish hospitals by asking patients referred to surgery: "What matters to you on the day of surgery"? This observational study has three goals:

1. To explore what matters to patients on the day of surgery
2. To explore associations between patients' degree-of-worry and their surgical fear on the day of surgery
3. To explore the characteristics and intensity of degree-of-worry

From 7.00 AM to 11.00 PM patients will be invited to answer:

1. What matters to them on the day of surgery and why it matters
2. How worried they are about their situation using a scale from 1 to 10, and to state why they worry.
3. Eight questions about their fear related to anesthesia and surgery on a scale from 0-10

In the analysis we will investigate the possible association between patients' degree of worry and fear related to anesthesia and surgery. Secondly, we analyse the prevalence of degree of worry and fear according to gender, age, type of surgery and medical speciality.

Finally, we will investigate what themes appear when we analyse the answers to what matters and why patients' worry.

ELIGIBILITY:
Inclusion Criteria:

* Danish speaking
* 18 years old or above

Exclusion Criteria:

* Patients who are not cognitively intact
* Do not consent to participation
* Patients requiring immediate surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish speaking adults referred to any type of planned surgery on June 6 2024
Sampling Method: Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Degree of worry | June 2024
  How worried are patients on the day of surgery on a scale from 1-10

SECONDARY OUTCOMES:
Surgical fear | June 2024
  How fearful are patients based on an 8-item scale with total score ranging from 0-80

OTHER OUTCOMES:
Agreement between degree of worry and surgical fear | 2024
  Measure of agreement using Cohen's kappa
What matters to you | 2025
  A thematic analysis of the answers to the question what matters to you
Integration of the qualitative and quantitative data | 2025
  Mixed methods analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hejdi Gamst-Jensen, SR, Study Director — Rigshospitalet, Denmark; Anne H Nielsen, Ass. prof., Study Chair — Gødstrup Hospital; Lone Brix, Lecturer, Study Director — University of Aarhus
Locations (1):
- Gødstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No